CLINICAL TRIAL: NCT02497716
Title: Single-dose Study Testing Rivaroxaban Granules for Oral Suspension Formulation in Children From 2 Months to 12 Years With Previous Thrombosis
Brief Title: Phase I Study on Rivaroxaban Granules for Oral Suspension Formulation in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17992; 2015-000962-76 (EudraCT Number)
Record Dates: First submitted 2015-07-12; First posted 2015-07-14 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rivaroxaban (Experimental): Single arm, open label study
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939 — Single dose of reconstituted rivaroxaban granules

SUMMARY:
To characterize the pharmacokinetic profile of rivaroxaban administered as granules for suspension formulation and to document safety and tolerability

ELIGIBILITY:
Inclusion Criteria:

* Children with an age ≥2 months and weight between 3 and <12 kg, who have completed anticoagulant treatment at least 10 days prior to the planned study drug administration.

  * Gestational age at birth of at least 37 weeks
  * Oral feeding/ nasogastric/ gastric feeding for at least 10 days
* Normal PT and aPTT within 10 days prior to planned study drug administration
* Written informed consent provided and, if applicable, child assent provided

Exclusion Criteria:

* Active bleeding or high risk for bleeding, contraindicating anticoagulant therapy
* Planned invasive procedures, including removal of central lines, within 24 hours before and after single dose intake
* An estimate glomerular filtration rate (eGFR) < 30 mL/min/1.73m2
* Hepatic disease which is associated either with:

  * coagulopathy leading to a clinically relevant bleeding risk, or alanine aminotransferase (ALT) > 5x upper level of normal (ULN), or
  * total bilirubin > 2x ULN with direct bilirubin > 20% of the total.
* Platelet count < 50 x 10^9/L
* Hypertension (defined as systolic and/or diastolic blood pressure >95th percentile for age)
* Concomitant use of strong inhibitors of both CYP3A4 and P-glycoprotein, e.g., all human immunodeficiency virus protease inhibitors and the following azoleantimycotic agents: ketoconazole, itraconazole, voriconazole, and posaconazole, if used systemically (fluconazole is allowed)
* Concomitant use of strong inducers of CYP3A4, e.g., rifampicin, rifabutin, phenobarbital, phenytoin and carbamazepine
* Inability to cooperate with the study procedures
* Hypersensitivity to rivaroxaban
* Participation in a study with an investigational drug other than rivaroxaban or a medical device within 30 days prior to treatment
* History of gastrointestinal disease or surgery associated with impaired absorption

Ages: 2 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

PRIMARY OUTCOMES:
AUC (area under the curve) | 4x within 8 hrs post study drug administrationh and 1x between 24-28h after administration
  Only PK will be tested in central lab
Cmax (maximum observed drug concentration) | 4x within 8 hrs post study drug administrationh and 1x between 24-28h after administration
  Only PK will be tested in central lab

SECONDARY OUTCOMES:
Prothrombin time (PT) | Pre-administration, if not done within the past 10 days, and then 24-28 hours after drug administration
Activated partial thromboplastin time (aPTT) | Pre-administration, if not done within the past 10 days, and then 24-28 hours after drug administration
Composite of major bleeding and clinically relevant non-major bleeding | From dose administration until follow up call on day 8+3

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (21):
- United States (5):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Oakland, Oakland, California
  - Riley Hospital For Children, Indianapolis, Indiana
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
- UZ Leuven Gasthuisberg, Leuven, Belgium
- Canada (4):
  - University of Alberta Hospital, Edmonton, Alberta
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
- Finland (2):
  - HUS Lastenklinikka, HUS
  - Turun yliopistollinen keskussairaala, kantasairaala, Turku
- France (2):
  - Hôpital Arnaud de Villeneuve - Montpellier, Montpellier
  - Hopital Necker les enfants malades - Paris, Paris
- University of Semmelweis/ Semmelweis Egyetem, Budapest, Hungary
- Italy (3):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - A.O.U. Città della Salute e della Scienza di Torino, Turin, Piedmont
  - A.O. di Padova, Padua, Veneto
- Spain (3):
  - Hospital de Sant Joan de Déu, Esplugues de Llobregat, Barcelona
  - Ciutat Sanitària i Universitaria de la Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid